CLINICAL TRIAL: NCT00000993
Title: An Open Protocol for the Use of Zidovudine for Prophylactic Treatment of Individuals After Accidental Massive Exposure to the Human Immunodeficiency Virus (HIV)
Brief Title: A Study of Zidovudine in the Prevention of HIV Infection in Individuals Exposed to the Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Prevention
Other Study IDs: NS 402
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 1991-04

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Evaluation; Accidents; Acquired Immunodeficiency Syndrome; AIDS Serodiagnosis; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To prevent individuals who have had a massive accidental exposure to HIV from becoming infected with HIV and possibly developing AIDS, by treating them with zidovudine (AZT). Although the number of persons who have been (or will be) exposed to a high concentration of HIV is quite small, these persons have a high risk of becoming infected and treatments are needed to prevent infection after such an exposure. In animal studies, AZT has prevented the development of infections after exposure of the animals to a retrovirus (the HIV is a retrovirus). In patients with AIDS, AZT has been effective in delaying the progression of the disease. For these reasons a trial of AZT is indicated.

DETAILED DESCRIPTION:
Although the number of persons who have been (or will be) exposed to a high concentration of HIV is quite small, these persons have a high risk of becoming infected and treatments are needed to prevent infection after such an exposure. In animal studies, AZT has prevented the development of infections after exposure of the animals to a retrovirus (the HIV is a retrovirus). In patients with AIDS, AZT has been effective in delaying the progression of the disease. For these reasons a trial of AZT is indicated.

Persons accepted into the study will take AZT capsules every 4 hours (6 times daily) for 42 days. Treatment with AZT should start as soon as possible, but no later than 5 days, after exposure to the HIV. Blood and urine samples for various studies will be taken at intervals during the 42-day treatment period, and blood samples will be taken every 3 months for 1 year and every 6 months for 2 years and tested for signs of HIV infection (HIV antibody determinations).

ELIGIBILITY:
Inclusion Criteria

Participant must be HIV-negative at entry and source must be HIV-positive. The source should be documented to be infected with HIV by one of the following criteria:

* Clinical diagnosis of AIDS or ARC.
* Positive test for HIV antibody (both ELISA and Western blot) or presence of HIV p24 antigen in serum.
* Participant may be enrolled if the source of exposure is suspected of being infected with HIV (member of risk group, some type of symptom of HIV infection), but the source must be confirmed to be infected with HIV for the participant to remain in the study.
* Significant exposure within 5 days prior to beginning therapy, defined as one of the following:
* Research laboratory workers or auxiliary personnel who, during the course of their work, were exposed to high titers of virus on abraded skin or mucous membranes or were accidentally inoculated with high titers of cell-associated or free virus through an exposed wound or puncture.
* Organ transplant recipients from HIV-positive donor.
* Recipients of blood or blood products from HIV-positive donor.
* Women who have been artificially inseminated with semen from HIV-positive donor.
* Other sources of exposure considered appropriate by the principal investigator and the sponsor.
* Persons with poor health (such as renal, hepatic, or bone marrow insufficiency) will be evaluated on a case-by-case basis.

Exclusion Criteria

Prior Medication:

Excluded within 4 weeks of study entry:

* Treatment with any potentially myelosuppressive drug.
* Nephrotoxic agents.
* Other experimental therapy.

Prior Treatment:

Excluded within 1 month of study entry:

* Blood transfusion with evidence of compromised blood marrow function.

Patients may not have any of the following:

* History of a malignancy other than cutaneous basal cell or cervical carcinomas.
* Significant, chronic underlying medical illness which, in the physician's judgment, would impair study completion.
* Liver dysfunction with bilirubin > 5 x ULN, alkaline phosphatase > 5 x upper limit of normal, or SGPT > 5 x upper limit of normal.
* Compromised bone marrow function with hemoglobin < 11 g/dl or blood transfusion within the last month, granulocytes < 1500 cells/mm3, or platelets < 100000/mm3.

When possible, no other concomitant medication will be administered during the treatment period.

Prior diagnosis of HIV infection by one of the following criteria:

* HIV antibody positive by ELISA or Western blot assays.
* HIV p24 antigen positive.
* Clinical symptoms which lead to a diagnosis by a licensed physician of AIDS / AIDS related complex (ARC) / AIDS dementia.

Active drug or alcohol abuse sufficient in the investigators' opinion to prevent compliance with the study regimen.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pettinelli C, Study Chair
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States